CLINICAL TRIAL: NCT02878681
Title: A 24-week, Randomized, Single-masked, Multicenter, Phase IV Study to Compare sysTemic VEGF Levels Following Monthly Intravitreal Injections of 0.5 mg Ranibizumab Versus 2 mg Aflibercept Until Week 24 in Patients With Visual Impairment DuE to Diabetic Macular Edema (TIDE DME).
Brief Title: 24 Week Study to Compare Systemic VEGF-levels of Ranibizumab and Aflibercept in DME.
Acronym: TIDE DME
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002D2404
Record Dates: First submitted 2016-07-22; First posted 2016-08-25 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Visual Impairment Due to Diabetic Macular Edema
Keywords: Diabetic Macular Edema.
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Monthly intravitreal injections of 0.5 mg ranibizumab for six months
  Interventions: Drug: Ranibizumab
- Group 2 (Experimental): Monthly intravitreal injections of 2 mg aflibercept for the initial three months followed by monthly intravitreal injections of 0.5 mg ranibizumab for the next three months.
  Interventions: Drug: Ranibizumab; Drug: Aflibercept
- Group 3 (Experimental): Monthly injections of 2 mg aflibercept for six months
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg intravitreal injections
  Other Names: Lucentis
  Arms: Group 1; Group 2
Drug: Aflibercept — 2 mg intravitreal injections
  Other Names: Eylea
  Arms: Group 2; Group 3

SUMMARY:
The purpose of the study is to compare the effect of intravitreal injections of ranibizumab and aflibercept on systemic VEGF levels in DME patients in a detailed time course.

DETAILED DESCRIPTION:
The purpose of the study is to compare the effect of monthly intravitreal injections of 0.5 mg ranibizumab and 2.0 mg aflibercept on systemic VEGF levels in patients with visual impairment due to DME over a 24 week period. In addition, the study will also assess the effect on systemic VEGF-A levels when patients are switched from aflibercept to ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Visual impairment due to DME
* BCVA of 78 to 24 (20/32-20/320) ETDRS letters

Exclusion Criteria:

* Stroke or myocardial infarction less than 3 months prior to screening.
* Presence of uncontrolled systolic blood pressure or diastolic blood pressure
* Renal failure requiring dialysis or renal transplant or renal insufficiency
* Untreated diabetes mellitus
* Use of any systemic anti-VEGF drugs within 6 months prior to screening.
* Use of systemic or inhaled corticosteroids for at least 30 consecutive days within 3 months prior to screening.
* Women who are pregnant or breast feeding or who are menstruating and capable of becoming pregnant* and not practicing a medically approved method of contraception

For either eye:

* Any active periocular or ocular infection or inflammation
* Uncontrolled glaucoma
* Neovascularization of the iris or neovascular glaucoma
* History of treatment with any anti-angiogenic drugs

For study eye:

* Atrophy or fibrosis involving the center of the fovea at the time of screening or baseline.
* Cataract (if causing significant visual impairment), planned cataract surgery during the study period, vitrectomy, aphakia, glaucoma surgery, severe vitreous hemorrhage, rhegm
* Irreversible structural damage within 0.5 disc diameter of the center of the macula
* Panretinal laser photocoagulation within 6 months prior to randomization.
* Focal/grid laser photocoagulation within 3 months prior to randomization.
* Any intraocular procedure (including cataract surgery, Yttrium-Aluminum-Garnet capsulotomy) within 3 months prior to baseline or anticipated within the next 6 months following
* Topical ocular corticosteroids administered for at least 30 consecutive days within 3 months prior to screening.
* Application of intravitreal corticosteroids in vitreous within 6 months prior to screening. Prior application of fluocinolonacetonid releasing implant in vitreous within 36 months prior to screening.

For fellow eye

- Retinal or choroidal neovascularization or macula edema of any cause Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of VEGF-A levels from baseline to week 24 | baseline to week 24
  Systemic VEGF-A levels following monthly intravitreal injections of 0.5 mg ranibizumab versus 2 mg aflibercept (Area under the curve) expressed in pg/ml*days. The AUC will be standardized (=divided) by the individual follow-up time and will be calculated by the trapezoidal rule..

SECONDARY OUTCOMES:
Mean Systemic VEGF-A levels in serum for patients in treatment group 1 and treatment group 2 within specific time points | Day 7, Day 15, Week 4, week 8, week 12, week 14, week 16, week 18, week 20, week 24
  To compare systemic VEGF-A levels (pg/ml) in patients switching from monthly 2 mg aflibercept injections for first three months to monthly 0.5 mg ranibizumab (treatment group 2) for the next three months compared to patients treated with monthly 0.5 mg ranibizumab (treatment group 1) for six months at specific time points from week 12 to week 24. The comparison will be performed at specific time points between week 12 and week 24, based on the blood samples collected for visits 10 to 16.
Mean Systemic VEGF-A levels in serum for patients in treatment group 1 and treatment group 3 within specific time points | Day 7, Day 15, Week 4, week 8, week 12, week 14, week 16, week 18, week 20, week 24
  To compare systemic VEGF-A levels (pg/ml) in patients switching from monthly 2 mg aflibercept injections for first three months to monthly 0.5 mg ranibizumab (treatment group 2) for the next three months compared to patients treated with monthly 2 mg aflibercept (treatment group 3) for six months at specific time points from week 12 to week 24. The comparison will be performed at specific time points between week 12 and week 24, based on the blood samples collected for visits 10 to 16.
Proportion of patients reporting ocular and/or systemic adverse events in all the three treatment groups. | From Baseline to Week 24
  To evaluate ocular and systemic safety in all the three treatment groups. Only treatment-emergent AEs will be summarized.
  AEs will be summarized by presenting for each treatment group the number and percentage of patients having any AE, having an eye-related AEs, having an AE in each primary system organ class and having each individual AEs based on the preferred term. All other information collected (e.g., severity or relationship to study treatment) will be tabulated and listed as appropriate. Summary tables will also be presented for the subset of AEs suspected to be treatment related.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals